CLINICAL TRIAL: NCT05554653
Title: Influence of Leucine Enriched Amino Acids on Myofibrillar and Collagen Protein Synthesis in Human Skeletal Muscle
Brief Title: Influence of Leucine Enriched Amino Acids on Myofibrillar and Collagen Protein Synthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daniel Moore (Other)
Responsible Party: Sponsor-Investigator, Daniel Moore, Associate Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ULE
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Interventional
Keywords: Leucine-enriched amino acids; Carbohydrate Placebo

STUDY DESIGN:
Intervention Model Description: Crossover to receive LEAA or Carbohydrate placebo. Unilateral leg exercise to give 4 outcome. (1) LEAA-EX; (2) LEAA-REST; (3) PLACEBO-EX; (4) PLACEBO-REST
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded (investigators and participants). A lab member external to the investigation will code items for the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leucine enriched essential amino acids (Active Comparator): Leucine enriched essential amino acids (4g total, of which 1.6g are leucine). 20g carbohydrate, 2g of protein free drink powder, and 5g of Splenda to mask taste.
  Interventions: Dietary Supplement: Leucine enriched amino acids
- Carbohdyrate Placebo (Placebo Comparator): Iso-caloric placebo (4g maltodextrin to replace LEAA). 20g carbohydrate, 2g of protein free drink powder, and 5g of Splenda to mask taste.
  Interventions: Dietary Supplement: Carbohydrate Placebo

INTERVENTIONS:
Dietary Supplement: Leucine enriched amino acids — Leucine enriched essential amino acids (4g total, of which 1.6g are leucine). 20g carbohydrate, 2g of protein free drink powder, and 5g of Splenda.
  Other Names: LEAA
  Arms: Leucine enriched essential amino acids
Dietary Supplement: Carbohydrate Placebo — iso-caloric placebo (4g maltodextrin). 20g carbohydrate, 2g of protein free drink powder, and 5g of Splenda.
  Arms: Carbohdyrate Placebo

SUMMARY:
The primary objective will be to determine the effect of leucine-enriched essential amino acids (LEAA) compared to carbohydrate placebo on dietary incorporation of [D5] Phenylalanine & [D5] Glycine into the three skeletal muscle protein pools (myofibrillar, sarcoplasmic and collagen), both following resistance exercise and at rest, with the two tracers provided as a 'intrinsically labeled' bolus. Other outcomes will relate to molecular regulation of protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male and female, recreationally-active participants.
* Healthy will be defined as screened by the PAR-Q+ (The Physical Activity Readiness Questionnaire for everyone; Appendix B).
* Self-reported not having engaged in resistance exercise and/or lower body plyometrics for at least 3 months prior to the study.
* Participants will be aged 18-35 years old.
* Participants are willing to abide by the compliance rules of this study.
* Self-reported regular menstrual cycle (25-35d) within the last 3 months (female participants).

Exclusion Criteria:

* Inability to adhere to any of the compliance rules judged by principle investigator or medical doctor.
* Self-reported regular tobacco use.
* Self-reported illicit drug use (e.g. growth hormone, testosterone, etc.).
* Individuals who have participated in studies within the past year involving any of the stable isotopes in the study.
* Use of birth control and discontinued use within the last 3 months (female participants).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar Protein synthesis | 4 hours
  Rate of incorporation of orally ingested amino acid tracers (D5 Phe and D5 Gly) into myofibrillar proteins isolated from skeletal muscle biopsies 4h following drink (LEAA or PLA) consumption and resistance exercise or at rest. Enrichment will be quantified via tandem LC-MS/MS to derive a rate of incorporation over the 4h period.

SECONDARY OUTCOMES:
Sarcoplasmic protein synthesis | 4 hours
  Rate of incorporation of orally ingested amino acid tracers (D5 Phe and D5 Gly) into sarcoplasmic (i.e., soluble) proteins isolated from skeletal muscle biopsies 4h following drink consumption (LEAA or PLA) and resistance exercise or at rest. Enrichment will be quantified via tandem LC-MS/MS.
Collagen protein synthesis | 4 hours
  Rate of incorporation of orally ingested amino acid tracers (D5 Phe and D5 Gly) into collagen (i.e., non-soluble) proteins isolated from skeletal muscle biopsies 4h following drink consumption (LEAA or PLA) and resistance exercise or at rest. Enrichment will be quantified via tandem LC-MS/MS.
Protein localization via immunofluorescence | 4 hours
  Antibody-determined Phosphorylated RPS6 (S240/244) and mTOR protein localization in human muscle cross sections and longitudinal sections as examined via immunofluorescence. Muscle sections (both longitudinal and cross-sections) will be derived from snap-frozen muscle biopsies performed 4h following drink consumption (LEAA or PLA) with or without resistance exercise (unilateral). Localization will be performed as done by Hodson et al., (2022; AJP Cell). Particularly, the localization of these targets relative to the cell periphery and z-discs (longitudinal sections only) will be analyzed via colocalization analysis.

OTHER OUTCOMES:
Isolation of primary myoblasts for in vitro nutritional experiments | 6-9 months
  isolation of primary myoblasts from skeletal muscle biopsies for growth in vitro and nutritional experiments in cell culture models

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada